CLINICAL TRIAL: NCT01923246
Title: Development of IVR and WEB Alcohol Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Claes Andersson, PhD, Region Skane
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: FHI 2006/100; 2006/100 (Other Grant/Funding Number: Swedish National Institute of Public Health)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Alcohol Consumption
Keywords: Alcohol consumption; Brief intervention; Automated techniques
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Single WEB intervention (Experimental): Web intervention recieved once.
  Interventions: Behavioral: Single WEB intervention
- Repeated WEB intervention (Experimental): Web intervention recieved twice.
  Interventions: Behavioral: Repeated WEB intervention
- Single IVR intervention (Experimental): IVR intervention recieved once
  Interventions: Behavioral: Single IVR intervention
- Repeated IVR intervention (Experimental): IVR intervention recieved twice
  Interventions: Behavioral: Repeated IVR intervention
- Control group (No Intervention): Untreated Control Group.

INTERVENTIONS:
Behavioral: Single WEB intervention — Brief WEB intervention recieved once
  Arms: Single WEB intervention
Behavioral: Repeated WEB intervention — WEB intervention recieved twice.
  Arms: Repeated WEB intervention
Behavioral: Single IVR intervention — IVR intervention recieved once
  Arms: Single IVR intervention
Behavioral: Repeated IVR intervention — IVR intervention recieved twice
  Arms: Repeated IVR intervention

SUMMARY:
The primary aim of the present study is to study the effect of a brief automated alcohol intervention in University students, and if there is a difference in effect between automated brief interventions delivered by internet (WEB) or Interactive Voice Response (IVR), and to study if there is difference in effect between single and repeated interventions.

ELIGIBILITY:
Inclusion Criteria:

* Females scoring 6 and above and males scoring 8 and above on AUDIT.

Exclusion Criteria:

* Females scoring 5 and below and males scoring 7 and below on AUDIT

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1672 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ALCOHOL USE DISORDERS IDENTIFICATION TEST (AUDIT) | September 2011 - October 2011

SECONDARY OUTCOMES:
Daily Drinking Questionnaire (DDQ) | September 2011 - October 2011

CONTACTS AND LOCATIONS:
Overall Officials: Claes Andersson, PhD, Principal Investigator — Malmö University, Department of Criminology
Locations (1):
- Malmö university, Department of Criminology, Malmo, Skåne County, Sweden